CLINICAL TRIAL: NCT05534841
Title: Assessment of Complete Response MRI Criterion After Neoadjuvant Therapy in Locally Advanced Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: 22.03.05
Record Dates: First submitted 2022-09-01; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Rectal Neoplasms
Keywords: MRI; Complete response
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pathological complete response: Patients with a complete response to the neoadjuvant therapy on the definitive anatomopathology study.
- Non pathological complete response: Patients without complete response to the neoadjuvant therapy on the definitive anatomopathology study.

SUMMARY:
Standard care for locally advanced rectal cancer consists in a neoadjuvant therapy followed by surgery. Morbidity and mortality remain high after rectal surgery, and often linked with quality of life impairment. 10 to 30% present a pathological complete response after neoadjuvant therapy. Some surgical teams propose "watch and wait" approach for patients selected with clinical complete responses criterion. The problem is to be sur the response is complete. MRI seems to be accurate to select complete responders. We will try to find MRI criterion of complete responses.

ELIGIBILITY:
Inclusion Criteria:

* Rectal adenocarcinoma
* Locally advanced
* Neoadjuvant therapy
* MRI restaging
* Rectal surgery
* Definitive anatomopathology study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Digestive surgery department
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-12 (Actual)

PRIMARY OUTCOMES:
Complete response MRI criterion | Day 0: immediately after the procedure
  We selected several objective MRI criterion among literature and compared them between the two groups.

SECONDARY OUTCOMES:
MRI accuracy | Day 0: immediately after the procedure
  Calculated Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Nîmes, Nîmes, GARD, France

IPD SHARING:
Plan to Share IPD: No